CLINICAL TRIAL: NCT02733718
Title: The Impact of Different Feeding Strategies During Packed Red Cell Transfusion on Intestinal Oxygenation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MR-01022016
Record Dates: First submitted 2016-02-28; First posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Necrotizing Enterocolitis
Keywords: Necrotizing enterocolitis; Transfusion; Mesenteric Oxygenisation
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: no enteral feeding (Other): intervention: NIRS (near-infrared spectroscopy)
  Interventions: Device: NIRS (near-infrared spectroscopy)
- Group 2: Feeding is reduced by %50 (Other): intervention: NIRS (near-infrared spectroscopy)
  Interventions: Device: NIRS (near-infrared spectroscopy)
- Group 3: Feeding will be continued (Other): intervention: NIRS (near-infrared spectroscopy)
  Interventions: Device: NIRS (near-infrared spectroscopy)

INTERVENTIONS:
Device: NIRS (near-infrared spectroscopy) — mesenteric oxygenisation measurement

SUMMARY:
This study aims to compare the differences between three different feeding regimens on intestinal oxygenation during packed red blood cell (PRBC) transfusion in premature babies.

DETAILED DESCRIPTION:
Necrotizing enterocolitis is an important cause of mortality and morbidity in neonates. Especially neonates, who are smaller than 32 weeks of gestational, need transfusions during their hospital stay. Recent evidences suggest a relation between antecedent PRBC transfusions and an increase in necrotizing enterocolitis (NEC). It has been reported that transfusion related NEC (TR-NEC) tend to occur immediately and up to 48 hours post-transfusion. Although the underlying mechanism of this relationship is still overinvestigation, altered oxygenation of the mesenteric vasculature during PRBC transfusion has been hypothesized to contribute to NEC development. But pathophysiology of this has not been cleared, yet. Nowadays, due to the increased risk of NEC during PRBC transfusion, different nutrition protocols are implemented in different units. These protocols contain permanent discontinuation, reducement or continuation of nutrition during the transfusion. As a result, there is still no evidence -based practice recommendation in this regard.

"Restricted Transfusion Guidelines" will be used for the decision of transfusion in premature infants. Patients will be divided into three different groups, according to their feeding regimen during transfusion.

Group 1: No enteral feeding before (two hours), during (3 hours) and after (two hours) red blood cell transfusion.

Group 2: Enteral feeding is reduced by %50 before, during and after the red blood cell transfusion.

Group 3: The same feeding volume will be continued without decreasing or stopping.

Groups will be determined with randomization. It was targeted to be at least twenty infants in each group. In all patients, mesenteric oxygenation will be compared before-during and after blood transfusion. Mesenteric oxygenation will be measured with Near Infrared Spectroscopy (NIRS), that is a non-invasive NIRS conducted technology. Cerebral oxygenation and peripheral oxygen saturations will be measured at the same timeline.

The investigators primary aim is to show the best method of feeding during transfusion that causes less feeding intolerance and NEC. The secondary outcomes will be the risk factors associated with feeding intolerance and NEC during PRBC transfusion, in premature babies.

ELIGIBILITY:
Inclusion Criteria:

* Prematurity (<32 completed weeks of gestation at birth)
* Need for PRBC transfusion
* Feeding at least 30ml/kg/day at the time of transfusion

Exclusion Criteria:

* Neonates previously diagnosed with gastrointestinal problems such as NEC, intestinal perforation or atresia.
* Infants receiving continuous feeds or less than 30ml/kg/day
* Major congenital or chromosomal abnormalities or infants unlikely to survive
* Intraventricular hemorrhage >Grade 3
* Hemodynamically significant patent ductus arteriosus
* Infants requiring vasopressor support
* Skin disruption precluding application of sensors

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
mesenteric oxygenisation (number of participants that has low mesenteric oxygenisation after transfusion) | 48 hours
  number of participants that has low mesenteric oxygenisation after transfusion

SECONDARY OUTCOMES:
Feeding intolerance (number of participants that has feeding intolerance after transfusion) | starting with transfusion until discharge, assessed up to 12 weeks
  number of participants that has feeding intolerance after transfusion
NEC (number of participants that has occurred transfusion related NEC) | starting with transfusion until discharge, assessed up to 12 weeks
  number of participants that has occurred transfusion related NEC

CONTACTS AND LOCATIONS:
Overall Officials: Hülya Selva Bilgen, MD, Study Director — professor
Locations (1):
- Marmara University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Marin T. Mesenteric perfusion pattern changes as the result of packed red blood cell transfusions in preterm infants. (Doctoral Dissertation). 2012. Retrieved from Emory Electronic Theses and Dissertations Repository. UMI number 3522333. [cited 2013 Feb 20]
- [Result] Marin T, Moore J, Kosmetatos N, Roback JD, Weiss P, Higgins M, McCauley L, Strickland OL, Josephson CD. Red blood cell transfusion-related necrotizing enterocolitis in very-low-birthweight infants: a near-infrared spectroscopy investigation. Transfusion. 2013 Nov;53(11):2650-8. doi: 10.1111/trf.12158. Epub 2013 Mar 11. PMID 23480548
- [Result] Bailey SM, Hendricks-Munoz KD, Mally P. Splanchnic-cerebral oxygenation ratio as a marker of preterm infant blood transfusion needs. Transfusion. 2012 Feb;52(2):252-60. doi: 10.1111/j.1537-2995.2011.03263.x. Epub 2011 Jul 25. PMID 21790634
- [Result] Stritzke AI, Smyth J, Synnes A, Lee SK, Shah PS. Transfusion-associated necrotising enterocolitis in neonates. Arch Dis Child Fetal Neonatal Ed. 2013 Jan;98(1):F10-4. doi: 10.1136/fetalneonatal-2011-301282. Epub 2012 Mar 23. PMID 22447991
- [Result] Christensen RD, Lambert DK, Henry E, Wiedmeier SE, Snow GL, Baer VL, Gerday E, Ilstrup S, Pysher TJ. Is "transfusion-associated necrotizing enterocolitis" an authentic pathogenic entity? Transfusion. 2010 May;50(5):1106-12. doi: 10.1111/j.1537-2995.2009.02542.x. Epub 2009 Dec 29. PMID 20051059